CLINICAL TRIAL: NCT04827342
Title: Feasibility and Functionality Test of Ada's DDSS Prototype, Exploring the Potential and Performance When Diagnosing Complex Cases of Dyspnea at the Emergency Department and Ward of Interna! Medicine of the University Hospital Basel
Brief Title: Feasibility and Functionality Test of Ada's DDSS Prototype
Acronym: Ada4dyspnoe
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Ada Health GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-00095; me19Eckstein3
Record Dates: First submitted 2021-03-26; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Dyspnea
Keywords: Ada DDSS prototype; Diagnostic Decision Support System (DDSS)
MeSH Terms: conditions — Dyspnea | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection in the Ada DDSS prototype — Entry of patients' data (medical history, symptoms and findings) in the Ada DDSS prototype. The tool then automatically creates a list of possible diagnostic suggestions based on the information, which are compared with the diagnoses of the attending physician.

SUMMARY:
This study is to explore with a feasibility and functionality test the potential of the Ada DDSS prototype with cases of dyspnea patients using the data collected at the Emergency Department (ED) and the ward of Internal medicine of the University Hospital Basel.

DETAILED DESCRIPTION:
This is an observational i.e. non-interventional, prospective feasibility study, which assesses, through observation, the potential, functionality and diagnostic performance of the Ada DDSS prototype in evaluating patients presenting with dyspnea as primary predominant complaint to the ED.

Once the consent form is signed, the Investigator documents patients' data, medical history, symptoms and findings with the Ada DDSS prototype. During the entire patient journey through the hospital (presentation at the ED through to admission in the ward of Internal Medicine) relevant information are collected and documented in the Ada DDSS prototype simultaneously to standard documentation by the medical staff.

Examination and treatment are carried out by the attending physician without being influenced or affected by the entry of data in the Ada DDSS prototype.

There is no intervention/change made to the usual care, and therefore neither an intervention patient group nor a control patient group. The "usual care" that each patient receives is the control comparison point for the performance of the Ada DDSS. The diagnoses proposed by the tool at different times (after triage in the emergency centre, when transferred to the ward and when discharged from the hospital) are then compared with those of the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Dyspnea as the main symptom when entering the emergency room
* Existence of written consent
* The patient is able to speak, understand and read German or English.

Exclusion Criteria:

* Inability or unwillingness to understand and comply with study procedures due to:
* Language problems
* Acute mental disorders
* Dementia
* Clinical instability (e..B. resuscitation treatment, non-invasive ventilation, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyspnoea who come to the emergency room of the University Hospital Basel and are to be transferred to the Internal Medicine Ward due to their illness
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Ada DDSS prototype | during hospital stay (presentation at the ED through to admission in the ward of Internal Medicine, in the average 1 week)
  Feasibility of the Ada DDSS prototype simultaneously to standard documentation by the medical staff.
Subjectively perceived benefit from using the Ada DDSS prototype | during hospital stay (presentation at the ED through to admission in the ward of Internal Medicine, in the average 1 week)
  Subjectively perceived benefit from using the Ada DDSS prototype (during patient journey in the hospital) assessed by a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Timiliotis J, Blumke B, Serfozo PD, Gilbert S, Ondresik M, Turk E, Hirsch MC, Eckstein J. A Novel Diagnostic Decision Support System for Medical Professionals: Prospective Feasibility Study. JMIR Form Res. 2022 Mar 24;6(3):e29943. doi: 10.2196/29943. PMID 35323125